CLINICAL TRIAL: NCT07122336
Title: Optimized Ablation of the Posterior Wall in Persistent Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Doctor Liu, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OAPWAF
Record Dates: First submitted 2025-07-17; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PVI group (Sham Comparator): PVI
  Interventions: Procedure: PVI
- PVI+ PWI group (Experimental): PVI+ PWI
  Interventions: Procedure: PVI; Procedure: PWI
- PVI+ PWI+EGM group (Experimental): PVI+ PWI+EGM
  Interventions: Procedure: PVI; Procedure: PWI; Procedure: EGM

INTERVENTIONS:
Procedure: PVI — PVI
Procedure: PWI — PWI
  Arms: PVI+ PWI group; PVI+ PWI+EGM group
Procedure: EGM — EGM
  Arms: PVI+ PWI+EGM group

SUMMARY:
The design of this study is an intervention, randomized, controlled study and contains three randomized groups：（1）PVI group；（2）PVI+PWI group;（3）PVI+PWI+EGM group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. First-time ablation for persistent atrial fibrillation (PsAF)
3. Persistent AF definition: Sustained episodes lasting ≥7 days but ≤3 years (including episodes requiring pharmacologic or electrical cardioversion after ≥7 days)
4. Symptomatic AF with intolerance to at least one antiarrhythmic drug (AAD)
5. Documented PsAF episode: At least one recorded PsAF episode within the last 2 years prior to enrollment, confirmed by: ECG,Holter monitorin, Loop recorder, Telemetry, Transtelephonic monitoring (TTM),Implantable device
6. Ability and willingness to provide written informed consent
7. Compliance with all study follow-up requirements

Exclusion Criteria:

1. Paroxysmal AF: Episodes lasting <7 days (or requiring pharmacologic/electrical cardioversion <7 days)
2. Long-standing persistent AF: Continuous AF duration >3 years
3. No prior attempt/pursuit of cardioversion or sinus rhythm maintenance
4. Contraindications to systemic anticoagulation
5. Pregnancy
6. Advanced renal or hepatic failure
7. Severe valvular heart disease or cyanotic congenital heart disease
8. Hypertrophic cardiomyopathy (HCM)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from any documented atrial arrhythmia - atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL) - of more than 30 seconds, excluding the initial 3 months blanking period, at a minimum of 12 months follow up after a single ablat | 12 months

SECONDARY OUTCOMES:
Freedom from AF after a single procedure without anti-arrhythmic medications (excludes the blanking period) at 12 months | 12 months
Freedom from any AT episodes lasting more than 30 seconds after the blanking period without AADs after a single procedure | 12 months
The atrial fibrillation burden among study groups at 12-month follow-up (excluding the initial 3-month blanking period) after 1 to 2 ablation procedures, with or without discontinuation of antiarrhythmic drugs. | 12 months
Freedom from any documented atrial arrhythmia episodes lasting >30 seconds at 12-month follow-up (excluding the initial 3-month blanking period) after 1 to 2 ablation procedures, with or without discontinuation of antiarrhythmic drugs (AADs) | 12 months
Freedom from any documented sustained atrial arrhythmia episodes lasting >7 days at 12-month follow-up (excluding the initial 3-month blanking period) after 1 to 2 ablation procedures, with or without antiarrhythmic drug therapy | 12 months
freedom from any documented symptomatic atrial fibrillation/flutter/tachycardia episodes (>30 seconds) after assessment of all ablation procedures at final follow-up, excluding the initial 3-month blanking period. | 12 months
Procedure time / Fluoroscopy time / ablation time | 12 months
Periprocedural complications, including stroke, pulmonary vein stenosis, cardiac perforation, esophageal injury, and mortality. | 12 months
Quality of life assessments during ≥12-month follow-up (AFEQT) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No